CLINICAL TRIAL: NCT05667025
Title: Comparison of the Effects of Cycling Functional Electrical Stimulation and Conservative Rehabilitation Therapy on the Functional Status and Muscle Characteristics of Stroke Patients
Brief Title: Comparison of the Effects of Cycling FES and Conservative Rehabilitation Therapy on Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Serdar Kilinc, Assistant Professor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AIBU-FTR-SK-05
Record Dates: First submitted 2022-12-19; First posted 2022-12-28 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Hemiplegia
MeSH Terms: conditions — Hemiplegia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conservative Rehabilitation (Active Comparator): Conservative Rehabilitation
  Interventions: Other: Conservative rehabilitation
- Cycling Functional Electrical Stimulation in addition to Conservative Rehabilitation (Active Comparator): Cycling Functional Electrical Stimulation in addition to Conservative Rehabilitation
  Interventions: Other: Conservative rehabilitation; Other: Cycling Functional Electrical Stimulation in addition to Conservative Rehabilitation

INTERVENTIONS:
Other: Conservative rehabilitation — Joint range of motion, strengthening, balance-coordination and stretching exercises included in the conservative physiotherapy program 5 days a week for a total of 6 weeks
Other: Cycling Functional Electrical Stimulation in addition to Conservative Rehabilitation — In addition to conservative treatment, cycling FES to the affected lower extremity for 20 minutes, 3 days a week for 4 weeks. During the treatment, the patient will be seated on a chair and her feet will be fixed to the pedal with velcro tape, and the comfort during the treatment will be provided with calf supports.
  Arms: Cycling Functional Electrical Stimulation in addition to Conservative Rehabilitation

SUMMARY:
Comparison of the effects of cycling functional electrical stimulation and conservative rehabilitation therapy on the functional status and muscle characteristics of stroke patients

DETAILED DESCRIPTION:
Stroke is the second leading cause of death worldwide and is a major contributor to disability. It is one of the developments related to bleeding as a result of occlusion of blood vessels in the brain with a clot or damage from the vessels.Loss of strength and motor coordination in the lower and upper extremities is the main cause of disability after stroke. Activities such as walking, standing, sitting and daily activities such as dressing, bathing and toilet are frequently affected and sensorimotor disorders are common.

Functional electrical stimulation (FES) is one of the methods used in treatment. FES provides muscle contraction and movement by electrical stimulation of motor neurons. It is applied by a controller through skin electrodes to induce contractions. The FES-evoked bike allows people with or without voluntary leg movement to pedal an exercise bike on a fixed system.

In this study, the investigators aimed to compare the treatment efficacy and changes in muscle characteristics of conservative treatment and cycling FES in stroke patients.

Demographic data of the patients and healthy volunteers will be recorded. Hemiplegic patients will be evaluated in terms of Barthel Index, Modified Ashworth Scale, Berg Balance Scale, Functional Ambulation Scale, Brunnstrom's Hemiplegia Recovery Stage, Fatigue Severity Scale, Fugl-Meyer Assessment, 6-Minute Walking Test, Muscle strength measurement, pennation angle and thickness measurement of the musculus rectus femoris muscle

ELIGIBILITY:
Inclusion Criteria:

* Patients must be between the ages of 21-85.
* The time elapsed after stroke must be between 3-60 months.
* Patients must have had cerebrovascular disease for the first time.
* Patients' Functional Ambulation Scale grade ≤ 4
* Patients must be able to sit unsupported for 30 minutes and walk 6 meters with support or device.
* Patients' mini mental test score ≥ 24

Exclusion Criteria:

* Patients with peripheral nerve injury in the lower extremity
* Patients with a pacemaker or a pacemaker.
* Patients with severe spasticity of the lower extremities
* Patients with a history of more than one cerebrovascular disease
* Patients with a history of lower extremity fractures in the last 6 months
* Patients diagnosed with Parkinson, Multiple Sclerosis
* Patients with unstable cardiac pathology
* Patients' mini mental test score ≤ 24

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale | Before Treatment
  The BBS is used to objectively determine a patient's ability to balance safely during a predetermined set of tasks. The scale comprises 14 items. Each item receives a score ranging from 0 to 4, which is a five-point rank scale with 0 indicating the lowest level of functioning and 4 indicating the highest level of functioning
Berg Balance Scale | 6 Week After Treatment
  The BBS is used to objectively determine a patient's ability to balance safely during a predetermined set of tasks. The scale comprises 14 items. Each item receives a score ranging from 0 to 4, which is a five-point rank scale with 0 indicating the lowest level of functioning and 4 indicating the highest level of functioning
Functional Ambulation Scale | Before Treatment
  Functional Ambulation Scale is a 6-point functional walking test that evaluates ambulation ability and determines the amount of human support required by patients while walking, regardless of whether they use a personal assistive device. A score of 0 indicates that the patient has a dysfunctional ambulation A score of 5 denotes independent ambulation on any surface.
Functional Ambulation Scale | 6 Week After Treatment
  Functional Ambulation Scale is a 6-point functional walking test that evaluates ambulation ability and determines the amount of human support required by patients while walking, regardless of whether they use a personal assistive device. A score of 0 indicates that the patient has a dysfunctional ambulation A score of 5 denotes independent ambulation on any surface.
Brunnstrom Stages | Before Treatment
  Brunnstrom stages is a scale used to assess motor recovery after a stroke, which is expressed using values between 1 and 6. The higher the value on this scale, the higher would be the recovery.
Brunnstrom Stages | 6 Week After Treatment
  Brunnstrom stages is a scale used to assess motor recovery after a stroke, which is expressed using values between 1 and 6. The higher the value on this scale, the higher would be the recovery.

SECONDARY OUTCOMES:
Barthel Index | Before Treatment
  The Barthel index is used to assess activities of daily living. It consists of 10 items: feeding, bathing, grooming, dressing, bowel, bladder, toilet use, transfers, mobility, stairs. Scores range from 0-100. A score of 100 represents complete independence, and a score of 0 represents complete dependence.
Barthel Index | 6 Week After Treatment
  The Barthel index is used to assess activities of daily living. It consists of 10 items: feeding, bathing, grooming, dressing, bowel, bladder, toilet use, transfers, mobility, stairs. Scores range from 0-100. A score of 100 represents complete independence, and a score of 0 represents complete dependence.
Modified Ashworth Scale | Before Treatment
  Spasticity in the shoulder will be evaluated according to the Modified Ashworth Scale (MAS). The Modified Ashworth Scale is a 6-point scale. Scores range from 0 to 4, where lower scores represent normal muscle tone and higher scores represent increased degree of spasticity.
Modified Ashworth Scale | 6 Week After Treatment
  Spasticity in the shoulder will be evaluated according to the Modified Ashworth Scale (MAS). The Modified Ashworth Scale is a 6-point scale. Scores range from 0 to 4, where lower scores represent normal muscle tone and higher scores represent increased degree of spasticity.
6 min walking test | Before Treatment
  It is used to evaluate the functional capacity of patients. The patient is asked to walk in a 30-meter corridor marked at 3-meter intervals. At the end of the test, the distance walked by the patient is recorded in meters.
6 min walking test | 6 Week After Treatment
  It is used to evaluate the functional capacity of patients. The patient is asked to walk in a 30-meter corridor marked at 3-meter intervals. At the end of the test, the distance walked by the patient is recorded in meters.
Fatigue Severity Scale | Before Treatment
  The scale consists of 9 questions that test the fatigue severity of the subjects in the last week. It is scored from 1 to 7. The result is found by the arithmetic mean. 4 or more indicates severe fatigue.
Fatigue Severity Scale | 6 Week After Treatment
  The scale consists of 9 questions that test the fatigue severity of the subjects in the last week. It is scored from 1 to 7. The result is found by the arithmetic mean. 4 or more indicates severe fatigue.
Rectus Femoris Muscle Thickness | Before Treatment
  The linear probe of the ultrasound will be placed transversely at the midpoint of the distance between the trochanter major and the lateral space of the knee joint, and muscle thickness will be measured without applying pressure.
Rectus Femoris Muscle Thickness | 6 Week After Treatment
  The linear probe of the ultrasound will be placed transversely at the midpoint of the distance between the trochanter major and the lateral space of the knee joint, and muscle thickness will be measured without applying pressure.
Pennate angle | Before Treatment
  Pennate angle can be defined as the angle of entry of muscle fibers into the aponeurosis. At the point where the rectus femoris muscle thickness is measured, the investigators will turn the ultrasound probe horizontally and measure the pennate angle formed by 3 different muscle fibers with the bottom fascia by goniometry and record the arithmetic average of these measurements.
Pennate angle | 6 Week After Treatment
  Pennate angle can be defined as the angle of entry of muscle fibers into the aponeurosis. At the point where the rectus femoris muscle thickness is measured, the investigators will turn the ultrasound probe horizontally and measure the pennate angle formed by 3 different muscle fibers with the bottom fascia by goniometry and record the arithmetic average of these measurements.
Muscle strength measurement: | Before Treatment
  Knee extensor and flexor muscle strength will be measured with a North Coast hydraulic hand dynamometer. During the measurements, the knee will be in 90 degrees flexion while the patient is in a sitting position, the dynamometer will be placed in front of the ankle and the patient will be asked to push the dynamometer with all his strength, 3 measurements will be made and the average will be recorded as isometric knee extensor muscle strength. In the same way, the dynamometer will be placed behind the ankle and the patient will be asked to push the dynamometer with all his strength, the average of the 3 measurements will be taken and recorded as isometric knee flexor muscle strength.
Muscle strength measurement: | 6 Week After Treatment
  Knee extensor and flexor muscle strength will be measured with a North Coast hydraulic hand dynamometer. During the measurements, the knee will be in 90 degrees flexion while the patient is in a sitting position, the dynamometer will be placed in front of the ankle and the patient will be asked to push the dynamometer with all his strength, 3 measurements will be made and the average will be recorded as isometric knee extensor muscle strength. In the same way, the dynamometer will be placed behind the ankle and the patient will be asked to push the dynamometer with all his strength, the average of the 3 measurements will be taken and recorded as isometric knee flexor muscle strength.
Fugl-Meyer Assessment for lower extremity | Before Treatment
  In the lower extremity motor subscale, reflex activity in supine and sitting positions, flexor synergy in supine position, extensor synergy in side-lying position, combined synergies in sitting, non-synergy movements in standing, normal reflexes in sitting position are examined. Each item is scored with a 3-point ordinal scale (0: unable at all, 1: partially able, 2: fully able). The maximum score is 28.
Fugl-Meyer Assessment for lower extremity | 6 Week After Treatment
  In the lower extremity motor subscale, reflex activity in supine and sitting positions, flexor synergy in supine position, extensor synergy in side-lying position, combined synergies in sitting, non-synergy movements in standing, normal reflexes in sitting position are examined. Each item is scored with a 3-point ordinal scale (0: unable at all, 1: partially able, 2: fully able). The maximum score is 28.

CONTACTS AND LOCATIONS:
Overall Officials: Serdar Kılınç, Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Abant Izzet Baysal University, Bolu, Turkey (Türkiye)